CLINICAL TRIAL: NCT03757195
Title: Augmentation of Maxillary Horizontal And Vertical Bone Deficiency Using Mineralized Plasmatic Matrix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, hany mostafa ahmed, Resident of Oral Surgery in Nahda University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-11-16
Record Dates: First submitted 2017-11-27; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Alveolar Ridge Abnormality of Maxilla
Keywords: Mineralized plasmatic matrix; sticky bone; plasma; autogeous fibrin glue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- augmentation by xenograft (Experimental): xenograft mixed with plasma extracted from blood
  Interventions: Procedure: Augmentation

INTERVENTIONS:
Procedure: Augmentation — combination product

SUMMARY:
A new technique of grafting introduce called Mineralized plasmatic matrix. This technique can be used in grafting in anterior zone giving a good results and bone substitution occur using allograft or xenograft.

The bone graft have a good consistency when it mixed with plasma give easy application, strength and stability of the graft. Also plasma rich with CGF (Cellular growth factors).

DETAILED DESCRIPTION:
Patients suffering from anterior maxillary vertical and horizontal bone loss will be treated using a xeno-graft mixed with the same patient plasma that extracted from his own blood during the operation this graft will be stabilized by collagen membrane and surgical tags.

Patients will be follow up for 6 months to measure amount of bone loss of the xeno-graft during this period post operative using C.B.C.T

ELIGIBILITY:
Inclusion Criteria:

* Age: from 20 to 40 years old
* no history of previous grafting.
* no History of previous implant placement
* Medically Free e.g no debilitating diseases

Exclusion Criteria:

* Smoker patients.
* Alcoholic patients
* Pregnant.
* Drug Abusers.
* Hypertensive , Diabetic, having Problems or disease in Kidney and/or liver.
* Thyroid Disease.
* Problem in Vit.D absorption or in calcitonin hormone secretion.
* History of blood transfusion or donating blood less than 4 months.
* Patient under Corticosteroid therapy.
* Neurologicaly unstable patients.
* History of radiotherapy or chemo-therapy.
* Patient undergo Spect C.T Scan less than 4 Months .

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-07-29 (Estimated); Study Completion 2020-10-25 (Estimated)

PRIMARY OUTCOMES:
amount of bone loss | change from baseline at 6 months
  amount of bone loss after xenograft by CBCT

CONTACTS AND LOCATIONS:
Overall Officials: Tarek I. Abdallah, P.H.D, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Cairo Univerisity, Cairo
  - Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: No